CLINICAL TRIAL: NCT02844257
Title: Transfusion Dependency at Diagnosis and Transfusion Intensity During Initial Chemotherapy Are Associated With Poorer Outcomes in Adult Acute Myeloid Leukaemia
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0464
Record Dates: First submitted 2016-07-20; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myeloid Leukaemia
Keywords: Acute myeloid leukaemia; Transfusion dependency; Transfusion intensity; Prognosis; Chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute myeloid leukaemia (AML) is a haematological malignant disease characterized by an uncontrolled proliferation of immature hematopoietic cells. Over the last two decades, clinical trials have demonstrated an improved response rate in younger adult AML. Aggressive induction plus more potent intensification programs with chemotherapy alone or chemotherapy plus stem cell transplantation (SCT) has improved treatment results. Advances in understanding disease biology, improvements in induction and consolidation program, and better supportive care have also all contributed. A number of clinical and laboratory characteristics influence the response to treatment and, thus, the survival of patients with AML. Among them, cytogenetic at diagnosis represents the most important prognostic variable. However, other factors may have a prognostic value and may influence patient's outcome.

Anaemia and thrombocytopenia are cardinal manifestations of AML. Over the last decades, it has become apparent that the frequency of allogeneic blood transfusions can modify host immunity and clinical outcomes. Anaemia has long been recognized as an adverse prognostic factor in myelodysplastic syndrome (MDS), which represents a pre-leukemic disease. Red blood cell (RBC) transfusion need was identified as a strong and independent risk factor for survival in MDS, for which the presence and severity of anaemia were attributed to a clonally advanced and biologically more aggressive disease.

Based on these data, the investigators retrospectively assessed the prognostic value of RBC and platelet transfusions at the time of diagnosis and the frequency of transfusions during the first induction course of chemotherapy in a large unselected group of patients with previously untreated AML.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 15 years old
* Newly diagnosed AML or post myelodysplastic syndrome (MDS)

Exclusion Criteria:

* Patients with M3 AML of French-American-British (FAB) classification (APL, Acute Promyelocytic Leukemia)
* World Health Organization (WHO) performance status >2; (ii)
* Left ventricular systolic ejection fraction below the normal range
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Serum creatinine concentration > 2x ULN (Upper Limit of Normal laboratory ranges),
* AST or ALT levels > 2.0 x upper limit of normal (ULN), except if AML-related

Ages: 15 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute myeloid leukaemia (AML)
Sampling Method: Non-Probability Sample
Enrollment: 1067 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Date of last contact if alive (up to 11 months)
  Overall survival (OS) is defined as the time elapsed between induction chemotherapy regimen and death for any cause. Patients not known to have this event are censored on the date they were last examined

SECONDARY OUTCOMES:
Complete remission (CR) rate | up to 11 months
  Response to induction therapy was assessed after one or two courses of chemotherapy (Between day 28 and day 35 of each course of chemotherapy). CR was defined according to standard criteria as less than 5 % blasts in bone marrow aspirates with evidence of maturation of cell lines and restoration of peripheral blood counts.
Number of blood products for each type of administration | Duration of study (11 months)
  Transfusion of a single unit of packed red blood cell (PRBC) or one whole-blood-derived platelet concentrate (PC) or platelets collected by apheresis (PA).
  Prophylactic transfusions were consistently given at morning platelet counts of <20×109/l and haemoglobin level <80 g/l. Patients requiring platelets were transfused with PC (PCs pooled from several units with 0.7 to 1×1011 platelets/10 kg of weight). Blood products were leukoreduced through discarding the buffy coat and administered through a standard blood filter but were not irradiated or routinely leukodepleted. Only patients planned to be allografted or autografted were transfused with irradiated transfusion products.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier THOMAS, MD-PhD, Principal Investigator — Hospices Civils de Lyon - Centre Hospitalier Lyon Sud
Locations (1):
- Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, 165 Chemin du Grand Revoyet, Pierre-Bénite, France